CLINICAL TRIAL: NCT04916249
Title: Tibetree Pain-Relieving Plaster for Musculoskeletal Pain Among Cancer Survivors
Brief Title: Testing an Herbal Pain Relief Patch to Reduce Pain in Cancer Survivors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-496
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Remission
Keywords: Tibetree; Tibetree Pain-Relieving; Cancer; Pain; Cancer survivor; 20-496; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Intervention Model Description: This is a single-center, two-arm, randomized, placebo-controlled trial comparing Tibetree PRP with a placebo control plaster.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study coordinators, patients, PI, co-investigators, biostatisticians will be blinded to which treatment group the patient was assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tibetree pain relieving plaster (Experimental): Participants with chronic musculoskeletal pain for ≥ 3 months and with BPI worst pain rated 5 or greater during the preceding week will be eligible for the study. We will enroll 66 participants with 33 patients in each arm.
  Interventions: Drug: Tibetree Pain Relieving Plaster
- Placebo plaster groups (Placebo Comparator): Participants with chronic musculoskeletal pain for ≥ 3 months and with BPI worst pain rated 5 or greater during the preceding week will be eligible for the study. We will enroll 66 participants with 33 patients in each arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tibetree Pain Relieving Plaster — Participants who provide informed consent in the trial will receive either the Tibetree pain relieving plaster if randomized into the intervention arm, or an identical placebo plaster if randomized into the control arm. The treatment course for both arms are identical. Participants will be instructed to apply the plaster directly to the skin overlying the area of pain for 6 hours once daily for 14 consecutive days.
  Other Names: Tibetree RP
  Arms: Tibetree pain relieving plaster
Other: Placebo — Participants who provide informed consent in the trial will receive either the Tibetree pain relieving plaster if randomized into the intervention arm, or an identical placebo plaster if randomized into the control arm. The treatment course for both arms are identical. Participants will be instructed to apply the plaster directly to the skin overlying the area of pain for 6 hours once daily for 14 consecutive days.
  Arms: Placebo plaster groups

SUMMARY:
The purpose of this study is to find out whether Tibetree Pain Relieving Plaster, an herbal pain relief patch, may be able to reduce this pain. Tibetree Pain Relieving Plaster is available as an over-the-counter (non-prescription) treatment for the temporary relief of minor aches and pains in muscles and joints. This study is the first to test this treatment in people who have had cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or older
* A diagnosis of cancer with no restrictions placed on type of cancer or stage. Eligibility criteria will not be restricted to MSK confirmed biopsy/diagnosis. Participating institution's testing is sufficient for other study sites
* Completed active treatment (surgery, chemotherapy, and/or radiotherapy) at least one month prior to study initiation (patients on continued hormone treatment or maintenance targeted therapies will not be excluded).
* Patients currently have no evidence of disease
* Ambulatory (Karnofsky functional score of ≥ 60)
* Having a focused location of regional musculoskeletal pain (e.g. joints, extremities, back, neck) that can be covered by one patch of PRP
* Worst pain score (numeric pain rating scale) 5 or above in the preceding week
* Pain for at least 3 months and at least 15 days with pain in the preceding 30 days; and willingness to adhere to and understanding of all study-related procedures, including randomization to one of the two possible choices
* Able to understand informed consent and provide signed informed consent form

Exclusion Criteria:

* Patients with non-musculoskeletal pain syndromes (headache, facial pain, chest pain, visceral abdominal pain) will be excluded if these are the sole source of pain but can be present as co-morbid conditions as long as a patient has a primary musculoskeletal pain condition defined as above.
* Patients have generalized musculoskeletal pain such as fibromyalgia
* Use of corticosteroid drugs by any route of administration within 30 days
* Patients with significant self-reported skin disorders
* Patients with open wounds, infections, skin trauma at skin overlying area of pain
* Patients with documented history of skin sensitivity to adhesive or allergic reaction to other patches or topical analgesics
* Patients with documented skin allergic reaction to plants or herbs
* Patients who are in active treatment (chemotherapy, surgery, radiotherapy)
* Plan to change or initiate other pain medications or interventions (e.g. physical therapy, acupuncture, injection). Patients may remain on their current pain regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2026-05-28 (Estimated); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory - Measure of Participant Pain | 14 days from baseline
  The short-form BPI will be used to quantify pain severity and pain interference. The BPI contains 4 pain severity items and 7 pain interference items, all rated on a scale from 0 to 10 (higher ratings indicate worse pain intensity/interference). A pain severity subscale score can be computed by taking the average rating of the 4 pain severity items. This subscale will be our primary outcome measure. A pain interference subscale score can be similarly computed for the 7 pain interference items. BPI should be completed prior to removing pain relieving plaster at the end of each day.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Mao, MD, MSCE, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk - Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Yang M, Baser RE, Li SQ, Hou YN, Chong K, Zhang YL, Hoque I, Bao T, Mao JJ. Tibetan Herbal Pain-Relieving Plaster for Chronic Musculoskeletal Pain Among Cancer Survivors: Study Protocol of a Randomized, Double-Blind, Placebo-Controlled Trial. Front Pharmacol. 2022 May 4;13:878371. doi: 10.3389/fphar.2022.878371. eCollection 2022. PMID 35600872
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org